CLINICAL TRIAL: NCT03885570
Title: Establishment of AI Prediction Model of Blood Transfusion Management in Patients With Mitral Valve Replacement
Brief Title: Blood Transfusion Management in Patients With Mitral Valve Replacement in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Qilu Hospital of Shandong University (Other); Zhejiang Provincial People's Hospital (Other); Beijing Aerospace General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ThirdXiangyaHCSUJF
Record Dates: First submitted 2019-01-30; First posted 2019-03-21 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-03

CONDITIONS: Mitral Valve Replacement; Transfusion Reaction; Blood Transfusion Complication
Keywords: mitral valve replacement; Predictive Model; Blood Transfusion; Perioperative period
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups/Cohorts: 1) Patients undergoing "mitral valve replacement" surgery;2) Age 18-75 years old;3) 48h preoperative biochemical indicators, blood general indicators, coagulation indicators are complete.
  Interventions: Procedure: Mitral valve replacement

INTERVENTIONS:
Procedure: Mitral valve replacement — Blood transfusion

SUMMARY:
The evaluation uses ΔHb as an independent factor combined with artificial intelligence (AI) to predict its impact on the prognosis and blood transfusion of patients undergoing cardiac surgery, thereby guiding perioperative clinical blood use and improving patient prognosis.

DETAILED DESCRIPTION:
1. Select 8 hospitals to form a multi-center team, and enter the keyword "mitral valve replacement" in the case system of 8 hospitals to collect information on 2000 heart surgery patients.
2. Mainly collect information on preoperative, intraoperative and postoperative test indexes (blood routine, liver and kidney function, coagulation function, blood gas), cardiac color Doppler, blood transfusion and prognosis of patients undergoing cardiac surgery, using statistical methods for analysis. Identify key observations.
3. Gradually incorporate and exclude data, and use statistical methods to conduct preliminary analysis on the collected data.

The AI prediction model was established by machine learning algorithm to predict intraoperative blood transfusion, verify the specificity and sensitivity of the blood transfusion prediction model, and scientifically guide clinical blood use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing "mitral valve replacement" surgery;
2. Age 18-75 years old;
3. 48h biochemical indicators before surgery, blood general indicators, coagulation indicators are complete.

Exclusion Criteria:

1. Lack of necessary tests and patient test information is not detailed, blood transfusion information is not detailed;
2. The blood transfusion information is not detailed in the same period as other cardiac operations (such as aortic valve surgery, coronary artery bypass grafting, etc.), but the tricuspid valvuloplasty is not ruled out at the same time;
3. Heart surgery or emergency surgery again.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with "mitral valve replacement" surgery who meet the standard in China, 18<Age<75.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2019-12-02 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 2 year
  The mortality during and after hospitalization
Intraoperative blood transfusion | through study completion, an average of 1 year
  The amount of intraoperative blood component input

CONTACTS AND LOCATIONS:
Overall Officials: Rong Gui, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- Third Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Schipper LJ, Baharoglu MI, Roos YBWEM, de Beer F. Medical Treatment for Spontaneous Anticoagulation-Related Intracerebral Hemorrhage in the Netherlands. J Stroke Cerebrovasc Dis. 2017 Jul;26(7):1427-1432. doi: 10.1016/j.jstrokecerebrovasdis.2017.03.019. Epub 2017 Apr 12. PMID 28412317
- [Background] Spolverato G, Bagante F, Weiss M, He J, Wolfgang CL, Johnston F, Makary MA, Yang W, Frank SM, Pawlik TM. Impact of Delta Hemoglobin on Provider Transfusion Practices and Post-operative Morbidity Among Patients Undergoing Liver and Pancreatic Surgery. J Gastrointest Surg. 2016 Dec;20(12):2010-2020. doi: 10.1007/s11605-016-3279-8. Epub 2016 Sep 30. PMID 27696209
- [Background] Spolverato G, Kim Y, Ejaz A, Frank SM, Pawlik TM. Effect of Relative Decrease in Blood Hemoglobin Concentrations on Postoperative Morbidity in Patients Who Undergo Major Gastrointestinal Surgery. JAMA Surg. 2015 Oct;150(10):949-56. doi: 10.1001/jamasurg.2015.1704. PMID 26222497
- [Background] Hogervorst E, Rosseel P, van der Bom J, Bentala M, Brand A, van der Meer N, van de Watering L. Tolerance of intraoperative hemoglobin decrease during cardiac surgery. Transfusion. 2014 Oct;54(10 Pt 2):2696-704. doi: 10.1111/trf.12654. Epub 2014 Apr 14. PMID 24724943
- [Background] Karkouti K, Wijeysundera DN, Yau TM, McCluskey SA, van Rensburg A, Beattie WS. The influence of baseline hemoglobin concentration on tolerance of anemia in cardiac surgery. Transfusion. 2008 Apr;48(4):666-72. doi: 10.1111/j.1537-2995.2007.01590.x. Epub 2008 Jan 10. PMID 18194382